CLINICAL TRIAL: NCT03573986
Title: Pilot Study of 18F-FMISO PET/CT and MRI Imaging to Explore Tissue Hypoxia and Arteriovenous Shunting in Subjects With Recurrent Glioblastoma Before and After Bevacizumab Treatment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 02318
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — fluoromisonidazole; Bevacizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Biological: [18F]fluoromisonidazole; Drug: Bevacizumab; Radiation: positron emission tomography (PET/CT).

INTERVENTIONS:
Biological: [18F]fluoromisonidazole — positron emitting radiopharmaceutical that has been studied in vivo in humans for measurement of regional hypoxia in a number of tumor types with positron emission tomography (PET/CT)
  Other Names: 18F-FMISO
Drug: Bevacizumab — Bevacizumab (Avastin, Genentech/Roche) is a humanized monoclonal antibody that binds to VEGF preventing its interaction with VEGFRs resulting in suppression of VEGF signaling.
Radiation: positron emission tomography (PET/CT). — PET-CT Scan 1.) before start of Bevacizumab up to approximately 4 weeks and 2.) within 12-22 days of start of Bevacizumab

SUMMARY:
Subjects with recurrent glioblastoma who are candidates for bevacizumab treatment according to standard of care will be eligible for this study. Positron emission tomography (PET/CT) imaging will use the investigational radiotracer [18F]FMISO to image the brain and evaluate for hypoxia pre and post therapy.. Subjects will also undergo up to three Brain MRIs.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥ 18 years of age
* Biopsy proven glioblastoma
* Must meet one of the following criteria:
* Recent surgery (within 2 months) showing recurrent glioblastoma with measurable (20 mm in 2 dimensions) residual tumor.

Radiologic evidence of recurrent tumor based on conventional and advanced MRI findings.

* Recommended for clinically indicated bevacizumab therapy
* Life expectancy of greater than 3 months in the opinion of an investigator or treating physician.
* Karnofsky performance status ≥ 60
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
* Less than 3 months from finishing the most recent radiation or immunotherapy.
* Contraindications to MRI or use of gadolinium contrast
* Only individuals (aged 18 or over) who can understand and give informed consent will be approached to participate in this study. Individuals who are considered to be mentally disabled will not be recruited for this study. All subjects must understand and be able to give informed consent. We will not be using specific methods to assess decisional capacity. Economically disadvantaged persons will not be vulnerable to undue influence, as this study offers no compensation. All individuals will be told that their choice regarding study participation will in no way change their access to clinical care. This should negate any undue influence or coercion. Pregnant women, children, fetuses, neonates, or prisoners are not included in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Ali Nabavizadeh, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States